CLINICAL TRIAL: NCT04064112
Title: Slanted Bilateral Lateral Rectus Recession Versus Conventional Bilateral Lateral Rectus Recession for Convergence Insufficiency Intermittent Exotropia in Children
Brief Title: S-BLR Versus C-BLR for CI-IXT in Children
Acronym: SCCIXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Zhao (Other)
Collaborators: Children's Hospital of Fudan University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Jiao Tong University School of Medicine (Other); Tianjin Eye Hospital (Other); Renmin Hospital of Wuhan University (Other); AIER Eye Hospital (Kunming) (Unknown)
Responsible Party: Sponsor-Investigator, Chen Zhao, Vice President of Department of Ophthalmology and Visual Science, Eye & ENT Hospital of Fudan University
Organization: Eye & ENT Hospital of Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019C-PEDIG
Record Dates: First submitted 2019-08-04; First posted 2019-08-21 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Convergence Insufficiency Intermittent Exotropia (CI-IXT)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-BLR (Experimental): For S-BLR, the lower horn of the LR is recessed based on near exodeviation and the upper horn is recessed based on distant exodeviation.
  Interventions: Procedure: S-BLR
- C-BLR (Active Comparator): For C-BLR, the LR is recessed based on distant exodeviation.
  Interventions: Procedure: C-BLR

INTERVENTIONS:
Procedure: S-BLR — Surgery of slanted bilateral LR recession for CI-IXT patients
  Arms: S-BLR
Procedure: C-BLR — Surgery of conventional bilateral lateral rectus recession for CI-IXT patients
  Arms: C-BLR

SUMMARY:
This is a multi-center, randomized single-blind controlled trial to compare the effectiveness of S-BLR with C-BLR for the treatment of CI-IXT in children.

Specific Aim 1 (Primary): To compare the surgical successful rate of S-BLR with C-BLR for the treatment of CI-IXT in children.

Specific Aim 2 (Secondary): To study the suboptimal surgical outcomes between S-BLR and C-BLR for the treatment of CI-IXT in children.

DETAILED DESCRIPTION:
Using conventional surgical procedures, higher postoperative near undercorrection and/or distant overcorrection rates were observed in CI-IXT. To achieve better outcome, S-BLR was introduced. Previous studies showed its efficacy in reducing near exodeviation, distant exodeviation, and NDD. So far, only limited studies have directly evaluated the surgical outcomes between S-BLR and C-BLR. The pilot study done by Snir et al included 12 patients with S-BLR and 6 patients with C-BLR and the success rates of S-BLR vs C-BLR were 92% vs 0 at one-year follow-up. The retrospective study done by Song et al included 17 patients undergoing S-BLR and 14 patients undergoing C-BLR. With stricter successful criteria, the success rates of S-BLR vs C-BLR were 35% vs 7% at six-month follow-up. A large randomized trial is needed to compare the surgical successful rate and suboptimal surgical outcomes of S-BLR with C-BLR in children with CI-IXT.

The proposed trial will be conducted in 6 different study sites working in the field of pediatric ophthalmology and strabismus.Each site will have one certified surgeon to do all surgeries. Under general anesthesia, the LR recession is performed using an inferior-temporal fornix incision. For S-BLR, the lower horn of the LR is recessed based on near exodeviation and the upper horn is recessed based on distant exodeviation. For C-BLR, the LR is recessed based on distant exodeviation. Surgical dose is according to the largest preoperative exodeviation at distance (6 meters) or near (1/3 meter) by the prism and alternate cover test(PACT). The extent of the recession is based on Parks' surgical dosage schedule.

ELIGIBILITY:
Inclusion Criteria:

* Exodeviation at least 15 at distance (6 meters);
* Exodeviation at most 50 at near (1/3 meter);
* Greater exodeviation at near than at distance by 10 or more;
* Control score of exodeviation greater than 3;
* Best-corrected visual acuity of 20/40 or better in the worse eye, and interocular difference of less than 2 lines;
* Myopia5.00D, hyperopia3.0D and anisometropia≤2.5D based on cycloplegic refraction
* Optical correction needed for at least 2 weeks before evaluation of exodeviation: myopia0.5D or astigmatism1.5D in either eye, or anisometropia1.0D;
* Written informed consent given by participants and their parents or legal guardians.

Exclusion Criteria:

* Prior strabismus surgery or botulinum toxin injection;
* Coexisting vertical deviation greater than 5, oblique muscle dysfunction, torsional deviation, dissociated vertical deviation, A-V pattern, or other conditions requiring horizontal rectus transposition, oblique surgery or vertical rectus surgery;
* Paralytic or restrictive strabismus;
* Lateral incomitance (greater exodeviation in right or left gaze position than in primary position by 5 or more with appropriate optical correction);
* Ocular disease other than strabismus or refractive error;
* Previous intraocular or refractive surgery;
* Craniofacial malformations affecting the orbit;
* Significant neurological disorders;
* Birth date34 weeks or birth weight1500 gram.

Abbreviations: CI-IXT, convergence insufficiency intermittent exotropia; D, diopter.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2022-02-19 (Actual); Study Completion 2023-02-11 (Actual)

PRIMARY OUTCOMES:
surgical successful rate | at 12 month
  Surgical successful cases/total cases. The successful criterion is a postoperative residual deviation at near and distance between 10 PD of exophoria/tropia and 5 PD of esophoria/tropia with near-distance difference <10 PD.

SECONDARY OUTCOMES:
suboptimal surgical rate | at 12 month
  suboptimal surgical cases/total cases. Suboptimal surgical outcomes include: undercorrection, overcorrection, diplopia, torsional deviation, A-V pattern, abduction limitation and reoperation.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Zhao, Doctor, Study Chair — Eye & ENT Hospital of Fudan University; Xiaoli Kang, Doctor, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University; Yueping Li, Doctor, Principal Investigator — Tianjin Eye Hospital; Lianhong Zhou, Doctor, Principal Investigator — Renmin Hospital of Wuhan University; Jing Yao, Doctor, Study Director — Eye & ENT Hospital of Fudan University; Chenhao Yang, Doctor, Principal Investigator — Children's Hospital of Fudan University; Jiangtao Xu, Doctor, Principal Investigator — AIER Eye Hospital (Kunming)
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
We concerns about patient privacy issues and it's better to protect the publication potential.

REFERENCES:
- [Background] Burian HM. Exodeviations: their classification, diagnosis and treatment. Am J Ophthalmol. 1966 Dec;62(6):1161-6. doi: 10.1016/0002-9394(66)92570-0. No abstract available. PMID 5957892
- [Background] Raab EL, Parks MM. Recession of the lateral recti. Effect of Preoperative fusion and distance-near relationship. Arch Ophthalmol. 1975 Aug;93(8):584-6. doi: 10.1001/archopht.1975.01010020568002. PMID 1156220
- [Background] Snir M, Axer-Siegel R, Shalev B, Sherf I, Yassur Y. Slanted lateral rectus recession for exotropia with convergence weakness. Ophthalmology. 1999 May;106(5):992-6. doi: 10.1016/S0161-6420(99)00522-9. PMID 10328402
- [Background] Chun BY, Kang KM. Early results of slanted recession of the lateral rectus muscle for intermittent exotropia with convergence insufficiency. J Ophthalmol. 2015;2015:380467. doi: 10.1155/2015/380467. Epub 2015 Jan 26. PMID 25688298
- [Background] Farid MF, Abdelbaset EA. Surgical outcomes of three different surgical techniques for treatment of convergence insufficiency intermittent exotropia. Eye (Lond). 2018 Apr;32(4):693-700. doi: 10.1038/eye.2017.259. Epub 2017 Dec 22. PMID 29271419
- [Background] Chen X, Fu Z, Yu J, Ding H, Bai J, Chen J, Gong Y, Zhu H, Yu R, Liu H. Prevalence of amblyopia and strabismus in Eastern China: results from screening of preschool children aged 36-72 months. Br J Ophthalmol. 2016 Apr;100(4):515-9. doi: 10.1136/bjophthalmol-2015-306999. Epub 2015 Aug 10. PMID 26261229
- [Background] Yang HK, Hwang JM. Surgical outcomes in convergence insufficiency-type exotropia. Ophthalmology. 2011 Aug;118(8):1512-7. doi: 10.1016/j.ophtha.2011.01.004. Epub 2011 Apr 7. PMID 21474185
- [Background] Wang B, Wang L, Wang Q, Ren M. Comparison of different surgery procedures for convergence insufficiency-type intermittent exotropia in children. Br J Ophthalmol. 2014 Oct;98(10):1409-13. doi: 10.1136/bjophthalmol-2013-304442. Epub 2014 May 19. PMID 24842862
- [Background] Ma L, Yang L, Li N. Bilateral lateral rectus muscle recession for the convergence insufficiency type of intermittent exotropia. J AAPOS. 2016 Jun;20(3):194-196.e1. doi: 10.1016/j.jaapos.2016.01.014. Epub 2016 May 6. PMID 27164428
- [Background] Choi DG, Rosenbaum AL. Medial rectus resection(s) with adjustable suture for intermittent exotropia of the convergence insufficiency type. J AAPOS. 2001 Feb;5(1):13-7. doi: 10.1067/mpa.2001.111137. PMID 11182666
- [Background] BURIAN HM, SPIVEY BE. THE SURGICAL MANAGEMENT OF EXODEVIATIONS. Am J Ophthalmol. 1965 Apr;59:603-20. No abstract available. PMID 14270998
- [Background] Kraft SP, Levin AV, Enzenauer RW. Unilateral surgery for exotropia with convergence weakness. J Pediatr Ophthalmol Strabismus. 1995 May-Jun;32(3):183-7. doi: 10.3928/0191-3913-19950501-12. PMID 7636700